CLINICAL TRIAL: NCT01382810
Title: A Randomized Masked Evaluation of Altaire Gel Forming Solution Versus Refresh Tears for the Treatment of Dry Eye Signs and Symptoms
Brief Title: Altaire Gel Forming Solution Versus Refresh Tears for the Treatment of Dry Eye Signs and Symptoms
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovative Medical (Industry)
Responsible Party: Melissa Earl, CRO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Altaire2011
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Dry Eye Syndromes
Keywords: dry eye signs and symptoms
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Altaire Gel forming solution (Active Comparator)
  Interventions: Drug: Altaire Gel forming solution
- Refresh Tears (Placebo Comparator)
  Interventions: Drug: Refresh Tears

INTERVENTIONS:
Drug: Altaire Gel forming solution — Three times a day for two months
  Arms: Altaire Gel forming solution
Drug: Refresh Tears — Three times a day for two months
  Arms: Refresh Tears

SUMMARY:
The purpose of this study is to evaluate and compare the effects of Altaire Gel forming solution and Refresh Tears in mild-moderate dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* Males or females.
* Patient reported dry eye symptoms (episodic, annoying, activity limiting).
* Physician assessment of mild-moderate dry eye.
* Patient willing to instill drops TID and complete entire length of protocol.
* TBUT _< 10 seconds.
* At least Grade 6 Corneal Staining.

Exclusion Criteria:

* Current topical cyclosporine use (Restasis)
* Current Refresh use.
* Refractive surgery within the last 6 months.
* Oral or topical corticosteroid use.
* Severe dry eye patients by physician assessment.
* Current active blepharitis.
* Oral doxycycline use.
* Oral antihistamine use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
TBUT | 2 months
  Test performed that measures how long the tears take to break up
Conjunctival and Corneal staining | 2 months
  Dye that will be placed inside the eye to evaluate the surface of the ey

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jackson Eye, SC, Lake Villa, Illinois
  - Koch Eye Associates, Warwick, Rhode Island